CLINICAL TRIAL: NCT01662531
Title: A Phase III Open-label, Multicenter, Pharmacokinetic, Safety and Efficacy Study of a Recombinant Fusion Protein Linking Coagulation Factor IX With Albumin (rIX-FP) in Previously Treated Children With Hemophilia B
Brief Title: A Safety, Efficacy and Pharmacokinetics Study of a Recombinant Fusion Protein Linking Coagulation Factor IX With Albumin (rIX-FP) in Children With Hemophilia B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSL654_3002; 2011-006032-23 (EudraCT Number)
Record Dates: First submitted 2012-08-07; First posted 2012-08-10 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — albutrepenonacog alfa

ARMS (1):
- rIX-FP (Experimental): Recombinant Fusion Protein Linking Coagulation Factor IX with Albumin (rIX-FP) will be administered by IV infusion as routine weekly prophylaxis and episodic treatment for bleeding episodes.
  Interventions: Biological: rIX-FP

INTERVENTIONS:
Biological: rIX-FP — Recombinant Fusion Protein Linking Coagulation Factor IX with Albumin (rIX-FP)

SUMMARY:
This study will examine the pharmacokinetics, safety and efficacy of rIX-FP for the control and prevention of bleeding episodes in children who have previously received factor replacement therapy for hemophilia B.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects, younger than 12 years old.
* Severe hemophilia B (Factor IX [FIX] activity of ≤ 2%).
* Body weight ≥ 10 kg.
* Subjects who have received FIX products (plasma-derived and/or recombinant FIX) for > 150 exposure days (EDs) (6 to < 12 years), and > 50 EDs (< 6 years).
* No history of FIX inhibitor formation, no detectable inhibitors at Screening and no family history of inhibitors against FIX.
* Written informed consent for study participation.

Exclusion Criteria:

* Known hypersensitivity to any FIX product or hamster protein.
* Known congenital or acquired coagulation disorder other than congenital FIX deficiency.
* Kidney or liver disease.
* Recent life-threatening bleeding episode.

Max Age: 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Study Director — CSL Behring
Locations (17):
- Australia (2):
  - The Royal Children's Hospital, Melbourne, Parkville, Victoria
  - The Children's Hospital at Westmead, Westmead
- AKH Wien (Paediatrics), Vienna, Austria
- McMaster Children's Hospital, Hamilton, Ontario, Canada
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Motole, Prague
- France (3):
  - C.R.T.H. Hopital de Bicentre (Hemophilie), Le Kremlin-Bicentre
  - Hospital Edouard Herriot, Lyon
  - Hôpital d'enfants La Timone, Marseille
- Germany (2):
  - CRC Coagulation Research Center GmbH, Duisburg/Altstadt
  - Universitätsklinikum Düsseldorf, Düsseldorf
- Sheba Medical Center, Tel Litwinsky, Israel
- Italy (2):
  - AOU Careggi, Florence
  - IRCCS Ospendale Maggiore (Centro emofilia e Trombosi), Milan
- FGU "Kirov Research Institute of Haemotology and Blood Trans), Kirov, Russia
- H.U. La Paz, Madrid, Spain

REFERENCES:
- [Derived] Alvarez-Roman MT, Merchan RD, Mellado RCR, Jimenez-Yuste V. Switching and increasing prophylaxis regimen with a genetically recombinant fusion of coagulation factor IX and albumin in haemophilia B: a case report. Curr Opin Hematol. 2023 Sep 1;30(5):175-179. doi: 10.1097/MOH.0000000000000775. PMID 37522479
- [Derived] Kenet G, Chambost H, Male C, Lambert T, Halimeh S, Chernova T, Mancuso ME, Curtin J, Voigt C, Li Y, Jacobs I, Santagostino E; PROLONG-9FP Investigator Study Group. Long-acting recombinant fusion protein linking coagulation factor IX with albumin (rIX-FP) in children. Results of a phase 3 trial. Thromb Haemost. 2016 Sep 27;116(4):659-68. doi: 10.1160/TH16-03-0179. Epub 2016 Sep 1. PMID 27583313

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 18 sites that were activated, subjects were enrolled from 17 sites in 10 countries.
Pre-assignment Details: Subjects <12 years of age with severe hemophilia B (FIX activity of ≤2%) were planned to be enrolled in the study, including 11 to 12 subjects in each age group (6 to <12 years and <6 years of age). Of 29 subjects screened, 27 subjects were enrolled and treated with rIX-FP.
Period: Overall Study
Arm/Group | rIX-FP
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All 27 subjects were included in the Safety, Pharmacokinetic and Efficacy populations.
Groups:
- Age < 6 Years: Subjects less than 6 years of age who received a single dose of 50 IU/kg rIX-FP on Day 1 during the pharmacokinetic phase of the study.
  Subjects received weekly (7-day) routine prophylaxis treatment with an initial weekly dose of 35 to 50 IU/kg rIX-FP, which may have been adjusted based on protocol-specified criteria.
- Age 6 to <12 Years: Subjects between 6 and less than 12 years of age who received a single dose of 50 IU/kg rIX-FP on Day 1 during the pharmacokinetic phase of the study.
  Subjects received weekly (7-day) routine prophylaxis treatment with an initial weekly dose of 35 to 50 IU/kg rIX-FP, which may have been adjusted based on protocol-specified criteria.
- Total: Total of all reporting groups
Arm/Group | Age < 6 Years | Age 6 to <12 Years | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.2 (1.70) | 8.1 (1.41) | 5.9 (2.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Incremental Recovery Following a Single Intravenous Dose of 50 IU/kg rIX-FP or Previous FIX Product
Description: Incremental recovery (IU/dL/IU/kg) is defined as the FIX activity (IU/dL) obtained 30 minutes following infusion, per dose of (IU/kg) infusion. FIX activity was measured at a central laboratory using validated one-stage clotting method. Recovery values were baseline-corrected for pre-infusion plasma FIX activity. Incremental recovery was measured following a single intravenous dose of 50 IU/kg rIX-FP on Day 1. Analysis of previous FIX product was conducted at the beginning of the study in a subset of subjects who had no historical pharmacokinetic (PK) data of their previous FIX product. For the PK assessment, the previous FIX product was administered by IV infusion after approximately 4 days following the last FIX treatment, prior to any dosing of rIX-FP. The formal PK population consisted of subjects who received at least 1 dose of rIX-FP for PK assessment and for whom a sufficient number of analyzable PK samples had been obtained to permit the evaluation of the PK profile of rIX-FP.
Time Frame: 30 minutes after infusion
Population: PK Population
Measure: Mean (Standard Deviation); unit: (IU/dL)/(IU/kg)
Groups:
- rIX-FP: All subjects received a single dose of 50 IU/kg rIX-FP on Day 1 during the pharmacokinetic phase of the study.
  Subjects received weekly (7-day) routine prophylaxis treatment with an initial weekly dose of 35 to 50 IU/kg rIX-FP, which may have been adjusted based on protocol-specified criteria.
Arm/Group | rIX-FP | Age < 6 Years | Age 6 to <12 Years
Number analyzed (Participants) | 27 | 12 | 15
(IU/dL)/(IU/kg)
  rIX-FP Assessment (n = 27, 12, 15) | 1.0114 (0.22711) | 0.9506 (0.20432) | 1.0600 (0.23934)
  Previous FIX Assessment (n = 17, 8, 9) | 0.7379 (0.19768) | 0.6764 (0.13980) | 0.7925 (0.23219)

2. Primary Outcome: Half-life (t1/2) Following a Single Intravenous Dose of 50 IU/kg rIX-FP or Previous FIX Product
Description: FIX activity was measured at a central laboratory using validated one-stage clotting method. FIX levels were not corrected for baseline values.
Time Frame: Pre-dose, 30 minutes, 3, 24, 48, 72 120, 168, 240 and 336 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | rIX-FP | Age < 6 Years | Age 6 to <12 Years
Number analyzed (Participants) | 27 | 12 | 15
hours
  rIX-FP Assessment (n = 26, 11, 15) | 91.4492 (15.9754) | 89.6124 (11.17364) | 92.7962 (19.02537)
  Previous FIX Assessment (n = 16, 7, 9) | 18.6291 (6.15551) | 19.8816 (8.01073) | 17.6550 (4.52497)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time Point Zero to the Last Sample With Quantifiable Drug Concentration (AUClast)
Description: AUClast following a single intravenous dose of 50 IU/kg rIX-FP or previous FIX product.
  FIX activity was measured at a central laboratory using validated one-stage clotting method. FIX levels were not corrected for baseline values.
Time Frame: Pre-dose, 30 minutes, 3, 24, 48, 72 120, 168, 240 and 336 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: IU*hr/dL
Arm/Group | rIX-FP | Age < 6 Years | Age 6 to <12 Years
Number analyzed (Participants) | 27 | 12 | 15
IU*hr/dL
  rIX-FP Assessment (n = 27, 12, 15) | 4156.7037 (1204.09549) | 3891.4820 (1252.99415) | 4368.8810 (1162.09967)
  Previous FIX Assessment (n = 16, 7, 9) | 718.9386 (230.52884) | 676.5414 (316.91381) | 751.9143 (146.70454)

4. Primary Outcome: Clearance for FIX Activity Following a Single Intravenous Dose of 50 IU/kg rIX-FP or Previous FIX Product
Description: FIX activity was measured at a central laboratory using validated one-stage clotting method. FIX levels were not corrected for baseline values. Clearance is normalized for body weight.
Time Frame: Pre-dose, 30 minutes, 3, 24, 48, 72 120, 168, 240 and 336 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | rIX-FP | Age < 6 Years | Age 6 to <12 Years
Number analyzed (Participants) | 27 | 12 | 15
mL/hr/kg
  rIX-FP Assessment (n = 26, 11, 15) | 1.1119 (0.31373) | 1.1841 (0.32924) | 1.0589 (0.30203)
  Previous FIX Assessment (n = 16, 7, 9) | 6.4007 (2.14434) | 7.1576 (2.78944) | 5.8119 (1.37641)

5. Primary Outcome: Number of Subjects Developing Inhibitors to Factor IX (FIX)
Description: Inhibitor formation was defined as any inhibitor (≥0.6 BU [Bethesda Units]/mL) identified and confirmed by retesting.
Time Frame: 12 months
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | rIX-FP
Number analyzed (Participants) | 27
participants | 0

6. Secondary Outcome: Number of Subjects With Treatment-related Adverse Events
Time Frame: 12 months
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | rIX-FP
Number analyzed (Participants) | 27
participants
  Any adverse event | 26
  Treatment-related adverse event | 0

7. Secondary Outcome: Number of Subjects Developing Antibodies Against rIX-FP
Description: Antibodies to rIX-FP were measured using a direct-binding enzyme-linked immunosorbent assay (ELISA).
Time Frame: 12 months
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | rIX-FP
Number analyzed (Participants) | 27
participants | 0

8. Secondary Outcome: Number of Bleeding Episodes Requiring One, Two or More Than Two Infusions of rIX-FP to Achieve Hemostasis
Description: For each bleeding episode that required treatment, the number of episodes that required one, two or more than two infusions of rIX-FP to achieve hemostasis
Time Frame: Approximately 12 months
Population: Efficacy Population
Measure: Number; unit: bleeding episodes
Arm/Group | rIX-FP | Age < 6 Years | Age 6 to <12 Years
Number analyzed (Participants) | 27 | 12 | 15
bleeding episodes
  1 infusion | 94 | 40 | 54
  2 infusions | 9 | 5 | 4
  > 2 infusions | 3 | 0 | 3
  1 or 2 infusions | 103 | 45 | 58

9. Secondary Outcome: Consumption of rIX-FP During Routine Prophylaxis
Description: Consumption of rIX-FP during routine prophylaxis is expressed as the total prophylaxis dose per month.
Time Frame: 12 months
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: IU/kg/month
Arm/Group | rIX-FP | Age < 6 Years | Age 6 to <12 Years
Number analyzed (Participants) | 27 | 12 | 15
IU/kg/month | 205.071 (41.1550) | 213.517 (44.3848) | 198.314 (38.5693)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Treatment-emergent adverse events, defined as adverse events present prior to the first dose of rIX-FP that subsequently worsened in severity or those that were not present prior to the first dose but subsequently appeared are summarized.
Arm/Group | rIX-FP
Serious Adverse Events (participants affected / at risk) | 4/27
Other Adverse Events (participants affected / at risk) | 23/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rIX-FP (N=27)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rIX-FP (N=27)
Contusion (Injury, poisoning and procedural complications) | 5 (9)
Injury (Injury, poisoning and procedural complications) | 2 (4)
Head injury (Injury, poisoning and procedural complications) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (4)
Pyrexia (General disorders) | 9 (14)
Dental discomfort (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (6)
Bronchitis (Infections and infestations) | 3 (4)
Ear infection (Infections and infestations) | 3 (4)
Gastroenteritis (Infections and infestations) | 3 (3)
Pharyngitis (Infections and infestations) | 2 (3)
Viral infection (Infections and infestations) | 2 (3)
Molluscum contagiosum (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.